CLINICAL TRIAL: NCT00911885
Title: A Simple Dietary Message to Improve Dietary Quality for Metabolic Syndrome
Acronym: CANDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Yunsheng Ma, Associate Professor, University of Massachusetts, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-13075
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Metabolic Syndrome
Keywords: Weight; Diet; Lipids
MeSH Terms: conditions — Metabolic Syndrome; Body Weight | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Fiber Diet (Experimental): A single dietary change condition that focuses exclusively on increasing fiber.
  Interventions: Behavioral: Dietary Intervention
- AHA Diet (Active Comparator): The AHA Diet is the current recommendation for patients with the metabolic syndrome.
  Interventions: Behavioral: Dietary Intervention

INTERVENTIONS:
Behavioral: Dietary Intervention — The efficacy of the two dietary change interventions will be compared in a randomized controlled trial, with 120 patients per group. The two approaches are 1) the American Heart Association (AHA) Dietary Guidelines; and 2) a simple dietary change condition that focuses on increasing fiber. Patients in both conditions will receive intensive dietary instruction for 3 months, followed by a 9 month maintenance phase. Both conditions will receive dietary instructions via individual and group sessions led by registered dietitians.

SUMMARY:
Identifying a simple dietary recommendation for weight loss and metabolic health may demonstrate potential for a simple public health message to impact coronary heart disease (CHD) prevention and metabolic syndrome. In a randomized clinical trial, the investigators propose to compare the efficacy of two intervention approaches to dietary change for CHD prevention among persons with metabolic syndrome. The two approaches are 1) the AHA Dietary Guidelines; and 2) a simple dietary change condition that focuses on increasing fiber. The investigators hypothesize that a message promoting high fiber intake may be the simple message that has potential to produce broad impact.

DETAILED DESCRIPTION:
The investigators will recruit 240 overweight and obese adults from a primary care setting who meet diagnostic criteria for metabolic syndrome. The efficacy of the two dietary change interventions will be compared in a randomized controlled trial, with 120 patients per group. The two approaches are 1) the American Heart Association (AHA) Dietary Guidelines; and 2) a simple dietary change condition that focuses on increasing fiber. Patients in both conditions will receive intensive dietary instruction for 3 months, followed by a 9 month maintenance phase. Both conditions will receive dietary instructions via individual and group sessions led by registered dietitians. Assessments, including diet, anthropometrics, blood pressure, fasting blood glucose, glycosylated hemoglobin (HbA1c), blood lipids, insulin, inflammatory markers, medication use, depression, quality of life, and physical activity will be conducted at baseline and at 6-, and 12-months after randomization. A 3-month post-intensive intervention assessment will measure short-term changes in body weight, diet, and metabolic syndrome indicators.

ELIGIBILITY:
Inclusion Criteria:

1. Meet diagnostic criteria for the metabolic syndrome;
2. Interested in losing weight and have a BMI 30-40.22 BMI>40 kg/m2 indicates severe obesity and is associated with functional limitations that are likely to prevent participation in the study;
3. Age 21 to 70 years old;
4. Telephone in the home or easy access to one;
5. Can provide informed consent;
6. Physician's approval to participate in the study;
7. Non-smoking status (given nicotine's effect on weight suppression, on HDL, and smoking cessation's effect weight gain); and
8. Ability to speak and read English.

Exclusion Criteria:

1. Has clinically diagnosed diabetes, or a fasting blood sugar of ≥ 126 mg/dl;
2. Had an acute coronary events within the previous 6 months;
3. Pregnant or lactating;
4. Women with polycystic ovary syndrome;133
5. Plans to move out of the area within the 12-month study period;
6. Diagnosis of a medical condition that precludes adherence to study dietary recommendations (e.g., Crohn's disease, ulcerative colitis, active diverticulitis, renal disease);
7. Has major depression or suicidality;
8. Is following a low-carbohydrate, high-fat dietary regimen such as the Atkins' Diet.134 Is participating in any current weight loss program;
9. Has had bariatric surgery or is currently using weight loss medication; and
10. Has an eating disorder (anorexia nervosa, bulimia nervosa or binge eating). Patients on lipid-lowering medications will not be excluded, but should be on a stable dose for 6 months.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2009-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Weight loss | 12 months

SECONDARY OUTCOMES:
Changes in components of the metabolic syndrome, inflammatory markers, LDL cholesterol, insulin levels, HbA1c, and diet | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yunsheng Ma, MD, Ph.D., Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Background] Olendzki BC, Ma Y, Schneider KL, Merriam P, Culver AL, Ockene IS, Pagoto S. A simple dietary message to improve dietary quality: Results from a pilot investigation. Nutrition. 2009 Jul-Aug;25(7-8):736-44. doi: 10.1016/j.nut.2009.01.009. Epub 2009 Apr 9. PMID 19359142
- [Background] Ma Y, Pagoto SL, Griffith JA, Merriam PA, Ockene IS, Hafner AR, Olendzki BC. A dietary quality comparison of popular weight-loss plans. J Am Diet Assoc. 2007 Oct;107(10):1786-91. doi: 10.1016/j.jada.2007.07.013. PMID 17904938
- [Background] Ma Y, Li W, Olendzki BC, Pagoto SL, Merriam PA, Chiriboga DE, Griffith JA, Bodenlos J, Wang Y, Ockene IS. Dietary quality 1 year after diagnosis of coronary heart disease. J Am Diet Assoc. 2008 Feb;108(2):240-6; discussion 246-7. doi: 10.1016/j.jada.2007.10.047. PMID 18237571
- [Background] Merriam PA, Ma Y, Olendzki BC, Schneider KL, Li W, Ockene IS, Pagoto SL. Design and methods for testing a simple dietary message to improve weight loss and dietary quality. BMC Med Res Methodol. 2009 Dec 30;9:87. doi: 10.1186/1471-2288-9-87. PMID 20042092
- [Background] Ma Y, Olendzki BC, Pagoto SL, Merriam PA, Ockene IS. What are patients actually eating: the dietary practices of cardiovascular disease patients. Curr Opin Cardiol. 2010 Sep;25(5):518-21. doi: 10.1097/HCO.0b013e32833cd538. PMID 20625282
- [Background] Wedick NM, Ma Y, Olendzki BC, Procter-Gray E, Cheng J, Kane KJ, Ockene IS, Pagoto SL, Land TG, Li W. Access to healthy food stores modifies effect of a dietary intervention. Am J Prev Med. 2015 Mar;48(3):309-17. doi: 10.1016/j.amepre.2014.08.020. Epub 2014 Oct 7. PMID 25300734
- [Background] Ma Y, Olendzki BC, Wang J, Persuitte GM, Li W, Fang H, Merriam PA, Wedick NM, Ockene IS, Culver AL, Schneider KL, Olendzki GF, Carmody J, Ge T, Zhang Z, Pagoto SL. Single-component versus multicomponent dietary goals for the metabolic syndrome: a randomized trial. Ann Intern Med. 2015 Feb 17;162(4):248-57. doi: 10.7326/M14-0611. PMID 25686165
- [Background] Wang J, Olendzki BC, Wedick NM, Persuitte GM, Culver AL, Li W, Merriam PA, Carmody J, Fang H, Zhang Z, Olendzki GF, Zheng L, Ma Y. Challenges in sodium intake reduction and meal consumption patterns among participants with metabolic syndrome in a dietary trial. Nutr J. 2013 Dec 18;12:163. doi: 10.1186/1475-2891-12-163. PMID 24345027
- [Background] Wang J, Persuitte G, Olendzki BC, Wedick NM, Zhang Z, Merriam PA, Fang H, Carmody J, Olendzki GF, Ma Y. Dietary magnesium intake improves insulin resistance among non-diabetic individuals with metabolic syndrome participating in a dietary trial. Nutrients. 2013 Sep 27;5(10):3910-9. doi: 10.3390/nu5103910. PMID 24084051
- [Background] Merriam PA, Persuitte G, Olendzki BC, Schneider K, Pagoto SL, Palken JL, Ockene IS, Ma Y. Dietary intervention targeting increased fiber consumption for metabolic syndrome. J Acad Nutr Diet. 2012 May;112(5):621-3. doi: 10.1016/j.jand.2012.01.024. Epub 2012 Apr 25. No abstract available. PMID 22709766
- [Derived] Zhang L, Pagoto S, May C, Olendzki B, L Tucker K, Ruiz C, Cao Y, Ma Y. Effect of AHA dietary counselling on added sugar intake among participants with metabolic syndrome. Eur J Nutr. 2018 Apr;57(3):1073-1082. doi: 10.1007/s00394-017-1390-6. Epub 2017 Mar 28. PMID 28353070